CLINICAL TRIAL: NCT03162068
Title: Specificities of Cushing's Osteoporosis Compare to Postmenopausal Osteoporosis : pQCT Analysis in Comparison With a Group of Controls.
Brief Title: Cushing's Osteoporosis Specificities
Acronym: SOCS
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Unité de recherche GReD CNRS UMR6293 / Inserm (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHU-334; 2016-A01482-49 (Other: 2016-A01482-49)
Record Dates: First submitted 2017-05-12; First posted 2017-05-22 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Osteoporosis in Cushing's Syndrome; Osteoporosis in Post-menopausal Women
Keywords: Cushing's syndrome; Osteoporosis; peripheral Quantitative Computed; volumetric Bone Mineral Density; Cortical and trabecular bone; Bone Strength
MeSH Terms: conditions — Cushing Syndrome; Osteoporosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control group: Cases are recruited thanks to advertisement within CHU.
  Interventions: Other: Osteodensitometry and pQCT
- Post menopausal women: Post-menopausal women are recruited within rheumatology service.
  Interventions: Other: Osteodensitometry and pQCT
- Cushing' syndrome group: Cushing' syndrome patients are recruited during hospitalisation in endocrinology service
  Interventions: Other: Osteodensitometry and pQCT

INTERVENTIONS:
Other: Osteodensitometry and pQCT — The peripheral Quantitative Computed analyses the bone architecture with distinction between cortical and trabecular compartment. We aim to determine the specificity of osteoporosis induced by glucocorticoids excess in comparison to post menopausal osteoporosis thanks to pQCT analysis.

SUMMARY:
Osteoporosis induced by glucocorticoids excess constitutes the main cause of secondary osteoporosis. Most of data available are provided from cohort studies of patients treated by corticosteroids, affecting among 1% of population. In contrast, very few data on osteoporosis are available in the Cushing syndrome (CS), a rare disease affecting 1 or 2 million of inhabitants, and characterized by an endogen glucocorticoid excess production. This affection is responsable of frequent fractures, occuring in 30-60% of patients (vertebral asymptomatic in 50% of case, hip, ribs). Fractures occurs often frequently above the threshold usually used for osteoporosis (T-score<-2.5), most often in the range of osteopenia. These data suggest that surface bone density isn't sufficient to characterize bone fragility, architectural factors are probably involved, and should be evaluated. The specificity of osteoporosis induced by endogen glucocorticoids excess in comparison with osteoporosis induced by estrogenic deficiency in post-menopausal women is poorly known, especially in endogen glucocorticoid excess.

A recent microarchitecture studies showed alterations of cortical compartment in patients with Cushing's syndrome, confirming by our preliminary preclinical data from a transgenic murin model of Cushing's syndrome.

In these ten last years, new radiologic tools have been developped, and are able to evaluate bone architecture. The peripheral Quantitative Computed analyses the bone architecture with distinction between cortical and trabecular compartment.

Therefore, we aim to determine the specificity of osteoporosis induced by glucocorticoids excess in comparison to post menopausal osteoporosis thanks to pQCT analysis.

DETAILED DESCRIPTION:
This study are divided in two parts :

- Cross sectional cohort with both comparison between : Cushing syndrome versus control and cushing syndrome versus post-menopausal women

Outcomes :

Primary outcomes : Analysis thanks to pQCT will be carried out in order to compare radius and tibia bone mineral volume (total, trabecular and cortical)

Secondary outcomes :

Strength parameters, muscle area adipose tissue surface will be assessed. Analysis of body composition thanks to DXA (Dual Energy X ray Absorptiometry), and surface bone mineral density.

Evaluation of Vertebral Fracture Assesment

- Prospective cohort with a longitudinal follow up on 5 years to assess the evolution of osteoporosis after treatment of Cushing syndrome (surgery or medical treatment).

CS patients are recruited during hospitalisation in endocrinology service Post-menopausal women are recruited within rheumatology service. Cases are recruited thanks to advertisement within CHU.

ELIGIBILITY:
Inclusion Criteria:

1. Cases

   * Healthy Volunteers
   * Men and women> 18 years
   * No known chronic treatment or pathology
   * Absence of tobacco or alcohol
   * Normal bone mineral density for age (Z-score> -2 and T-score> -2.5) and markers of bone remodeling in normal values for age and menopausal status (osteocalcin, CTX)
   * Free 24-hour urinary cortisol (CLU / 24 h) normal Cushing matching by menopausal status, age group, BMI, sex
2. Postmenopausal women

   * Menopause confirmed by hormonal assays
   * Amenorrhea for more than one year
   * Free 24-hour urinary cortisol (CLU / 24 h) normal
   * Osteoporosis confirmed at DXA (T score ≤ -2.5 DS) Post menopausal women matching according to BMI, T-DXA score (T score ≤ -2.5 DS)
3. Cushing's syndrome

   * Endogenous hypercorticism, whatever the cause (dependent or independent ACTH)
   * Active or controlled for less than 5 years

Exclusion Criteria:

1. Diseases with bone resonance:

   * Disease that can affect phosphocalcium metabolism or promote bone loss: endocrine diseases (hyperparathyroidism, hyperthyroidism); Osteomalacia, malabsorptive intestinal or inflammatory or chronic liver diseases, chronic inflammatory rheumatism.
   * Heavy comorbidities: heart failure or chronic respiratory insufficiency, known severe renal insufficiency.
2. Treatments:

   * Anti-osteoporotic treatments (bisphosphonates, raloxifene, denosumab)
   * Teriparatide; Lithium, thiazide diuretic, treatment with levothyrox suppressive dose, hormone replacement therapy of menopause, anticonvulsants, corticotherapy in progress or in the previous 5 years, anti-aromatases, anti-androgenic
3. Other:

   * Minors, pregnant women
   * Patients unable to express their will (sub-tutelage, curators, dementia).
   * Lack of social security
   * Lack of follow-up
   * Excessive consumption of alcohol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cushing syndrome group (CS): both Menopausal women Control: both
  Control = 24 Post menopausal women = 24 Cushing'syndrome group : n = 12
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2025-03-13 (Actual); Study Completion 2025-03-13 (Actual)

PRIMARY OUTCOMES:
Comparison of volumetric bone mineral density | at day 1
  thanks to pQCT with evaluation of total, trabecular and cortical compartment, between patients affecting by cushing'syndrome and post-menopausal women

SECONDARY OUTCOMES:
Assessment of strength bone of radius and tibia of the non-dominant limb | at day 1
  comparison Cushing syndrome versus both menopause women and controls : pQCT analysis
Assessment of trabecular and cortical compartment | at day 1
  comparison Cushing syndrome versus both menopause women and controls : pQCT analysis
Comparison of muscle area and surface, adipose tissue | at day 1
  comparison Cushing syndrome versus both menopause women and controls : pQCT analysis

CONTACTS AND LOCATIONS:
Overall Officials: Marie BATISSE-LIGNIER, Principal Investigator — CHU de Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, Auvergne, France